CLINICAL TRIAL: NCT03001115
Title: Post-Marketing Surveillance of Adalimumab in Korean Hidradenitis Suppurativa Patients Under the "New-Drug Re-examination
Brief Title: Post-Marketing Surveillance of Adalimumab in Korean Hidradenitis Suppurativa Subjects
Acronym: HS rPMS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-052
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Adalimumab; Safety; Hidradenitis Suppurativa; Korean participants
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Hidradenitis suppurativa (HS): Participants with HS treated with adalimumab (HUMIRA®) in routine clinical practice.

SUMMARY:
The objective of this study is to evaluate the safety profile of Adalimumab for Hidradenitis Suppurativa (HS) participants in normal medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participant who are eligible to be treated with adalimumab for HS in accordance with the approved Korean label
* Participant must provide written authorization form to use their personal health data prior to the participating in the study.

Exclusion Criteria:

* Participant who are contraindications to adalimumab as listed on the approved Korean label.
* Participant who is participating on other clinical trials.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hidradenitis suppurativa (HS) participants who have been prescribed Adalimumab by the treating investigator as per approved label in Korea will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Assessing adverse events | Up to 70 days following the last administration of Humira®
  Adverse event information is collected to assess prevalence of safety.

SECONDARY OUTCOMES:
Change from baseline in Dermatology Life Quality Index (DLQI) | Week 0 (baseline), Week 12, and Week 24
  DLQI will be collected to evaluate effectiveness of adalimumab. DLQI has 10 quality of life domains scored from 0 (no effect) to thirty (very large effect).
Change from baseline in Hidradenitis Suppurativa Clinical Response (HiSCR) | Week 0 (baseline), Week 12, and Week 24
  The HiSCR measure is designed to assess treatment response in a binary manner, rather than being a continuous or ordinal scale. It includes a count of the total number of abscesses and inflammatory nodules (ANs), as well as recording the number of sinuses draining purulent fluid present in an individual. Treatment responders are defined as those who achieve at least a 50% reduction in ANs, with no increase in the number of abscesses or draining sinuses, relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (19):
- South Korea (19):
  - Kyungpook National Univ Hosp /ID# 162930, Daegu, Daegu Gwang Yeogsi
  - Seoul National Univ Bundang ho /ID# 202254, Seongnam, Gyeonggido
  - CHA Bundang Medical center, CHA University /ID# 203364, Seongnam-si, Gyeonggido
  - Ajou University Hospital /ID# 163243, Suwon, Gyeonggido
  - Chonnam National University Hospital /ID# 162932, Gwangju, Jeonranamdo
  - Yonsei University Health System, Severance Hospital /ID# 162933, Seodaemun-gu, Seoul Teugbyeolsi
  - Seoul SongDo Hospital /ID# 202597, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital /ID# 162924, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 162934, Seoul, Seoul Teugbyeolsi
  - St. Mary's Hospital of the Cat /ID# 162923, Seoul, Seoul Teugbyeolsi
  - Dong-A University Hospital /ID# 162931, Busan
  - Korea University Anam Hospital /ID# 162922, Seoul
  - Seoul National University Hospital /ID# 162935, Seoul
  - Hangyang University Medical Ce /ID# 162929, Seoul
  - Konkuk University Medical Cent /ID# 162927, Seoul
  - Asan Medical Center /ID# 162925, Seoul
  - Hallym University Kangnam Sacred Heart Hospital /ID# 162926, Seoul
  - Ewha Womans University Mokdong /ID# 162928, Seoul
  - National Medical Center /ID# 162936, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P16-052.pdf